CLINICAL TRIAL: NCT05278000
Title: Improving Adherence to Controller Medication in Children With Asthma - the Unexplored Contribution of Behavioural Sciences
Brief Title: Improving Adherence to Controller Medication in Children With Asthma
Acronym: PACIFI
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Olivier Drouin, M.D., M.Sc M.P.H., Pediatrician and Clinical Assistant Professor, Departments of Paediatrics and Department of Social and Preventive Medicine, St. Justine's Hospital
Other Study IDs: 461392
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Asthma in Children; Adherence, Medication
Keywords: Asthma, Adherence, social needs, scarcity, future discounting
MeSH Terms: conditions — Medication Adherence; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children aged 2-17 years with asthma: Parents of children aged 2-17 years seen at CHU Sainte-Justine asthma clinic with a diagnosis of asthma will be eligible for the study
  Interventions: Other: Presence of scarcity mindset

INTERVENTIONS:
Other: Presence of scarcity mindset — This observational study will examine whether
  1. Individuals exhibiting a scarcity mindset have lower adherence to asthma controller medication
  2. Individuals with higher rates of future discounting have lower adherence to controller medication
  3. Individuals with unmet social needs are more likely to experience scarcity and have higher rates of future discounting, and whether these relationships mediate adherence to asthma controller medication
  Other Names: Presence of unmet social needs,; Rate of future discounting

SUMMARY:
Asthma is a common pediatric condition that can be well controlled with regular use of controller medications, however adherence to these is low, resulting in preventable exacerbations and important short- and long-term morbidity. This project's aim is to understand cognitive factors influencing adherence to medication among children with asthma, examining specifically the influence of scarcity (a mindset experienced by those with less than they need, which is cognitively taxing) and future discounting (the focus on present concerns at the expense of distant ones).

Using a single-centre, 12-month, prospective observation cohort study of 300 families of children with asthma, the objectives of this study are to:

1. Identify the relationship between scarcity, future discounting, and adherence to asthma medication.
2. Evaluate whether unmet social needs are associated with scarcity and future discounting.
3. Determine whether scarcity and future discounting mediate the relationship between unmet social needs and adherence to medication.

Primary outcome will be adherence to controller medication, which will be measured for the 12 months of follow-up on a scale of 0 to 100%, by the 'proportion of prescribed days covered (PPDC)', a validated index calculated as the number of days for which the drug was dispensed by a pharmacy, divided by the number of days for which it was prescribed. Other measures include screening families for unmet social needs, psychometric testing to document scarcity and future discounting.

This study will increase our understanding of how cognitive factors influence adherence to asthma controller medication, which will be instrumental in developing targeted interventions to improve adherence, especially for families experiencing with unmet social needs.

DETAILED DESCRIPTION:
Background: Asthma affects one in ten children and is among the most common causes of emergency department (ED) visits and hospitalization in paediatrics. Regular use of asthma controller medications is effective at controlling the condition, yet adherence to medication is low, resulting in preventable exacerbations and important short- and long-term morbidity. Higher adherence to asthma controller medications leads to more favourable health trajectories. Behavioural reasons for poor medication adherence may include cognitive mechanisms, such as scarcity (a mindset experienced by those with less than they need, which is cognitively taxing), and future discounting (the focus on present concerns at the expense of distant ones). Children living with socioeconomic disadvantage suffer a disproportionate burden of disease and are more likely to have unmet social needs such as food insecurity and unstable housing, leading to scarcity and future discounting.

Specific Objectives: This project's aim is to understand cognitive factors influencing adherence to medication among children with asthma, examining specifically the influence of scarcity and future discounting. Our objectives are to:

1. Identify the relationship between scarcity, future discounting, and adherence to asthma medication.
2. Evaluate whether unmet social needs are associated with scarcity and future discounting.
3. Determine whether scarcity and future discounting mediate the relationship between unmet social needs and adherence to medication.

Design: A single-centre, 24-month, prospective observational cohort study of 300 families of children with asthma. Follow-up includes two data collection time points at 6- and 12-months after recruitment.

Primary outcome will be adherence to controller medication, which will be measured for the 12 months of follow-up on a scale of 0 to 100%, by the 'proportion of prescribed days covered (PPDC)', a validated index calculated as the number of days for which the drug was dispensed by a pharmacy, divided by the number of days for which it was prescribed.

Other measures include: screening families for unmet social needs, psychometric testing to document scarcity and future discounting.

Relevance: This study will increase our knowledge of cognitive factors influencing adherence to asthma controller medication and will be instrumental in developing targeted interventions to improve adherence, especially for families experiencing with unmet social needs.

ELIGIBILITY:
Inclusion Criteria:

* (1) child with documented prescription for a controller medication at recruitment visit: inhaled corticosteroids ± Long-acting beta agonists (LABA) and/or Leukotriene receptor antagonists (LTRA)
* (2) consent to reMED database (medication data registry)

Exclusion Criteria:

* (1) Child with other chronic pulmonary disease (e.g., cystic fibrosis) that could influence asthma control,
* (2) parents' insufficient knowledge of French or English to complete questionnaires either alone or with support from a research assistant.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 300 families of children aged 2-17 who are followed at the CHU Sainte-Justine asthma or pulmonology clinic with a diagnosis of asthma (made according to national guidelines) and have a documented prescription for a controller medication at recruitment visit: inhaled corticosteroids ± Long-acting beta agonists (LABA) and/or Leukotriene receptor antagonists (LTRA)
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to controller medication | 12 months of follow up
  Measured on a scale of 0 to 100% by the proportion of prescribed days covered (PPDC), a well-validated index calculated as the number of days for which the drug was dispensed by a pharmacy, divided by the number of days for which it was prescribed. The PPDC will be calculated using data from the medical records and a medication database, reMED.

SECONDARY OUTCOMES:
Number of emergency room visits and/or hospitalizations related to asthma | 12 months of follow up
  Number of emergency room visits and/or hospitalizations related to asthma per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Drouin, MD, MSc MPH, Principal Investigator — CHU Sainte-Justine Research Centre, Université de Montréal
Locations (1):
- Asthma Clinic of the CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drouin O, Perez T, Barnett TA, Ducharme FM, Fleegler E, Garg A, Lavoie K, Li P, Metras ME, Sultan S, Tse SM, Zhao J. Impact of Unmet Social Needs, Scarcity, and Future Discounting on Adherence to Treatment in Children With Asthma: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2023 Mar 7;12:e37318. doi: 10.2196/37318. PMID 36881458